CLINICAL TRIAL: NCT02632409
Title: A Phase 3 Randomized, Double-blind, Multi-center Study of Adjuvant Nivolumab Versus Placebo in Subjects With High Risk Invasive Urothelial Carcinoma (CheckMate 274: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 274)
Brief Title: An Investigational Immuno-therapy Study of Nivolumab, Compared to Placebo, in Patients With Bladder or Upper Urinary Tract Cancer, Following Surgery to Remove the Cancer
Acronym: CheckMate 274
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA209-274; 2014-003626-40 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Various Advanced Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental): Nivolumab dose as specified
  Interventions: Biological: Nivolumab
- Placebo (Placebo Comparator): Placebo dose as specified
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Nivolumab
  Arms: Nivolumab
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of Nivolumab compared to placebo in participants who have undergone radical surgery for invasive urothelial cancer.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have had invasive urothelial cancer at high risk of recurrence originating in the bladder, ureter, or renal pelvis
* Must have had radical surgical resection (e.g. radical cystectomy), performed within the last 120 days
* Must have disease free status as determined by imaging within 4 weeks of dosing
* Tumor tissue must be provided for biomarker analysis
* Patients who have not received prior neoadjuvant cisplatin chemotherapy must be ineligible for or refuse cisplatin-based adjuvant chemotherapy

Exclusion Criteria:

* Partial bladder or partial kidney removal (eg, partial cystectomy or partial nephrectomy)
* Secondary Treatment (eg, adjuvant systemic chemotherapy for bladder cancer) following surgical removal of bladder cancer
* Subjects with active, known or suspected autoimmune disease
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured
* Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 day of study drug administration
* Positive test for hepatitis B virus surface antigen (HBV s Ag) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2027-05-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (188):
- United States (33):
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - Local Institution - 0179, Tucson, Arizona
  - Local Institution - 0061, Clovis, California
  - Local Institution - 0172, Sacramento, California
  - Local Institution - 0005, San Francisco, California
  - Local Institution - 0178, Lakewood, Colorado
  - Local Institution - 0167, Gainesville, Florida
  - Local Institution - 0030, Miami Beach, Florida
  - Local Institution - 0008, Tampa, Florida
  - Local Institution - 0168, Maywood, Illinois
  - Local Institution - 0094, Fort Wayne, Indiana
  - Local Institution - 0171, New Orleans, Louisiana
  - Local Institution - 0173, Grand Rapids, Michigan
  - Local Institution - 0051, Burnsville, Minnesota
  - Local Institution - 0004, Rochester, Minnesota
  - Local Institution - 0003, Omaha, Nebraska
  - Local Institution - 0177, Las Vegas, Nevada
  - Local Institution - 0176, Albany, New York
  - Local Institution - 0157, Buffalo, New York
  - Local Institution - 0007, Mineola, New York
  - Local Institution - 0001, New York, New York
  - Local Institution - 0006, New York, New York
  - Local Institution - 0166, Chapel Hill, North Carolina
  - Local Institution, Durham, North Carolina
  - Local Institution - 0044, Portland, Oregon
  - Local Institution - 0010, Portland, Oregon
  - Local Institution - 0180, Tigard, Oregon
  - Local Institution - 0074, Allentown, Pennsylvania
  - Local Institution - 0011, Pittsburgh, Pennsylvania
  - Local Institution - 0040, Pittsburgh, Pennsylvania
  - Local Institution - 0169, Myrtle Beach, South Carolina
  - Local Institution - 0009, Chattanooga, Tennessee
  - Local Institution - 0234, Norfolk, Virginia
- Argentina (6):
  - Local Institution - 0021, Berazategui, Buenos Aires
  - Local Institution - 0090, Capital Federal, Buenos Aires
  - Local Institution - 0089, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution - 0022, Ciudad Autónoma de BuenosAires, Buenos Aires
  - Local Institution - 0020, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0102, Viedma
- Australia (6):
  - Local Institution - 0048, Liverpool, New South Wales
  - Local Institution - 0047, St Leonards, New South Wales
  - Local Institution - 0046, Waratah, New South Wales
  - Local Institution - 0050, Elizabeth Vale, South Australia
  - Local Institution - 0184, Frankston, Victoria
  - Local Institution - 0175, Perth, Western Australia
- Austria (4):
  - Local Institution - 0133, Linz
  - Local Institution - 0136, Salzburg
  - Local Institution - 0132, Vienna
  - Local Institution - 0183, Vienna
- Belgium (2):
  - Local Institution - 0029, Hasselt
  - Local Institution - 0027, Liège
- Brazil (6):
  - Local Institution - 0071, Ijuí, Rio Grande do Sul
  - Local Institution - 0072, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0070, Barretos, São Paulo
  - Local Institution - 0073, Cerqueira César, São Paulo
  - Local Institution - 0231, Rio de Janeiro
  - Local Institution - 0100, São Paulo
- Canada (4):
  - Local Institution - 0139, Edmonton, Alberta
  - Local Institution - 0101, Montreal, Quebec
  - Local Institution - 0109, Montreal, Quebec
  - Local Institution - 0112, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0038, Viña del Mar, Región de Valparaíso
  - Local Institution - 0099, Santiago, Santiago Metropolitan
  - Local Institution - 0137, Temuco
- China (23):
  - Local Institution - 0191, Beijing, Beijing Municipality
  - Local Institution - 0206, Beijing, Beijing Municipality
  - Local Institution - 0192, Beijing, Beijing Municipality
  - Local Institution - 0210, Chongqing, Chongqing Municipality
  - Local Institution - 0198, Fuzhou, Fujian
  - Local Institution - 0222, Guangzhou, Guangdong
  - Local Institution - 0203, Guangzhou, Guangdong
  - Local Institution - 0227, Nanning, Guangxi
  - Local Institution - 0196, Wuhan, Hubei
  - Local Institution - 0220, Nanjing, Jiangsu
  - Local Institution - 0204, Nanjing, Jiangsu
  - Local Institution - 0223, Nanchang, Jiangxi
  - Local Institution, Xi'an, Shan3xi
  - Local Institution - 0212, Yantai, Shandong
  - Local Institution - 0193, Shanghai, Shanghai Municipality
  - Local Institution - 0202, Shanghai, Shanghai Municipality
  - Local Institution - 0199, Shanghai, Shanghai Municipality
  - Local Institution - 0217, Shanghai, Shanghai Municipality
  - Local Institution - 0229, Chengdu, Sichuan
  - Local Institution - 0219, Chengdu, Sichuan
  - Local Institution - 0221, Hangzhou, Zhejiang
  - Local Institution - 0195, Hangzhou, Zhejiang
  - Local Institution - 0230, Wenzhou, Zhejiang
- Colombia (3):
  - Local Institution - 0092, Bogotá
  - Local Institution - 0093, Floridablanca
  - Local Institution - 0091, Medellín
- Denmark (3):
  - Local Institution - 0108, Aalborg
  - Local Institution - 0106, Aarhus N
  - Local Institution - 0107, Copenhagen
- France (7):
  - Local Institution - 0233, Clermont-Ferrand
  - Local Institution - 0115, La Roche-sur-Yon
  - Local Institution - 0080, Marseille
  - Local Institution - 0081, Paris
  - Local Institution - 0113, Strasbourg
  - Local Institution - 0097, Suresnes
  - Local Institution - 0098, Villejuif
- Germany (12):
  - Local Institution - 0131, Chemnitz
  - Local Institution - 0125, Essen
  - Local Institution - 0127, Greifswald
  - Local Institution - 0126, Hamburg
  - Local Institution - 0124, Heidelberg
  - Local Institution - 0123, Jena
  - Local Institution - 0188, Marburg
  - Local Institution - 0122, Munich
  - Local Institution - 0128, Münster
  - Local Institution - 0185, Nuremberg
  - Local Institution - 0130, Regensburg
  - Local Institution - 0129, Stuttgart
- Greece (2):
  - Local Institution - 0110, Athens
  - Local Institution - 0111, Thessaloniki
- Ireland (2):
  - Local Institution - 0054, Wilton, CORK
  - Local Institution - 0052, Dublin
- Israel (4):
  - Local Institution - 0118, Haifa
  - Local Institution - 0121, Jerusalem
  - Local Institution - 0120, Ramat Gan
  - Local Institution - 0119, Ẕerifin
- Italy (8):
  - Local Institution - 0088, Arezzo
  - Local Institution - 0197, Bergamo
  - Local Institution - 0082, Milan
  - Local Institution - 0084, Pisa
  - Local Institution - 0189, Reggio Emilia
  - Local Institution - 0085, Roma
  - Local Institution - 0086, Roma
  - Local Institution - 0083, Siena
- Japan (16):
  - Local Institution - 0142, Akita, Akita
  - Local Institution - 0144, Hirosaki, Aomori
  - Local Institution - 0162, Fukuoka, Fukuoka
  - Local Institution - 0160, Sapporo, Hokkaido
  - Local Institution - 0161, Sapporo, Hokkaido
  - Local Institution - 0148, Tsukuba, Ibaraki
  - Local Institution - 0163, Nagasaki, Nagasaki
  - Local Institution - 0150, Niigata, Niigata
  - Local Institution - 0141, Okayama, Okayama-ken
  - Local Institution - 0149, Sayama, Osaka
  - Local Institution - 0151, Hamamatasu, Shizuoka
  - Local Institution - 0146, Bunkyo-ku, Tokyo
  - Local Institution - 0145, Shinjuku-Ku, Tokyo
  - Local Institution - 0147, Shinjuku-ku, Tokyo
  - Local Institution - 0143, Chiba
  - Local Institution - 0164, Osaka
- Mexico (6):
  - Local Institution - 0035, Guadalajara, Jalisco
  - Local Institution - 0138, Df, Mexico City
  - Local Institution - 0034, Mexico City, Mexico City
  - Local Institution - 0032, Monterrey, Nuevo León
  - Local Institution - 0116, México
  - Local Institution - 0039, México
- Netherlands (3):
  - Local Institution - 0069, Amsterdam, North Holland
  - Local Institution - 0068, Maastrict
  - Local Institution - 0041, Nijmegen
- Local Institution - 0043, Lima, Peru
- Poland (5):
  - Local Institution - 0055, Gdansk
  - Local Institution - 0057, Lodz
  - Local Institution - 0187, Warsaw
  - Local Institution - 0058, Wroclaw
  - Local Institution - 0186, Wroclaw
- Romania (4):
  - Local Institution - 0182, Bucharest
  - Local Institution - 0096, Craiova
  - Local Institution - 0078, Floreşti
  - Local Institution - 0181, Timisoara, Timis
- Russia (2):
  - Local Institution - 0140, Moscow
  - Local Institution - 0031, Saint Petersburg
- South Korea (4):
  - Local Institution - 0155, Seongnam-si
  - Local Institution - 0154, Seoul
  - Local Institution - 0152, Seoul
  - Local Institution - 0156, Seoul
- Spain (7):
  - Local Institution - 0067, Badalona-barcelona
  - Local Institution - 0066, Barcelona
  - Local Institution - 0064, Madrid
  - Local Institution - 0062, Madrid
  - Local Institution - 0063, Madrid
  - Local Institution - 0232, Santander
  - Local Institution - 0065, Seville
- Local Institution - 0105, Lund, Sweden
- Switzerland (2):
  - Local Institution - 0134, Basel
  - Local Institution - 0135, Zurich
- Taiwan (3):
  - Local Institution - 0158, Kaohsiung City
  - Local Institution - 0159, Taichung
  - Local Institution - 0153, Taipei
- United Kingdom (6):
  - Local Institution - 0025, Manchester, Greater Manchester
  - Local Institution - 0076, Edinburgh, Midlothian
  - Local Institution - 0024, Sutton, Surrey
  - Local Institution - 0059, Sheffield, Yorkshire
  - Local Institution - 0036, London
  - Local Institution - 0114, London

REFERENCES:
- [Derived] Galsky MD, Bajorin DF, Tomita Y, Ye D, Agerbaek M, Enting D, Peer A, Milowsky M, Kobayashi K, Grimm MO, Stenner F, David JM, Li J, Chasalow SD, Nasroulah F, Apfel A, Unsal-Kacmaz K, Necchi A. Adjuvant nivolumab in muscle-invasive urothelial carcinoma: exploratory biomarker analysis of the randomized phase 3 CheckMate 274 trial. Nat Med. 2025 Sep;31(9):3062-3073. doi: 10.1038/s41591-025-03802-8. Epub 2025 Aug 7. PMID 40775055
- [Derived] Geynisman DM, Chepynoga K, Yates G, Tate A, Kurt M, Patel MY, Teitsson S, Mitra S, Mamtani R. Estimating the Impact of Adjuvant Treatment With Nivolumab on Long-Term Survivorship Rates Compared With Surveillance in Muscle Invasive Urothelial Carcinoma: Mixture Cure Modeling Analyses of Disease-Free Survival From the Phase 3 CheckMate 274 Trial. Clin Genitourin Cancer. 2025 Jun;23(3):102335. doi: 10.1016/j.clgc.2025.102335. Epub 2025 Mar 17. PMID 40204616
- [Derived] Galsky MD, Witjes JA, Gschwend JE, Milowsky MI, Schenker M, Valderrama BP, Tomita Y, Bamias A, Lebret T, Shariat SF, Park SH, Agerbaek M, Jha G, Stenner F, Ye D, Giudici F, Dutta S, Askelson M, Nasroulah F, Zhang J, Brophy L, Bajorin DF. Adjuvant Nivolumab in High-Risk Muscle-Invasive Urothelial Carcinoma: Expanded Efficacy From CheckMate 274. J Clin Oncol. 2025 Jan;43(1):15-21. doi: 10.1200/JCO.24.00340. Epub 2024 Oct 11. PMID 39393026
- [Derived] Bajorin DF, Witjes JA, Gschwend JE, Schenker M, Valderrama BP, Tomita Y, Bamias A, Lebret T, Shariat SF, Park SH, Ye D, Agerbaek M, Enting D, McDermott R, Gajate P, Peer A, Milowsky MI, Nosov A, Antonio JN Jr, Tupikowski K, Toms L, Fischer BS, Qureshi A, Collette S, Unsal-Kacmaz K, Broughton E, Zardavas D, Koon HB, Galsky MD. Treatment of muscle-invasive urothelial cancer with nivolumab (CheckMate 274 study): a plain language summary. Future Oncol. 2023 Feb;19(6):413-426. doi: 10.2217/fon-2022-1294. Epub 2023 Mar 15. PMID 36919916
- [Derived] Witjes JA, Galsky MD, Gschwend JE, Broughton E, Braverman J, Nasroulah F, Maira-Arce M, Ye X, Shi L, Guo S, Hamilton M, Bajorin DF. Health-related Quality of Life with Adjuvant Nivolumab After Radical Resection for High-risk Muscle-invasive Urothelial Carcinoma: Results from the Phase 3 CheckMate 274 Trial. Eur Urol Oncol. 2022 Oct;5(5):553-563. doi: 10.1016/j.euo.2022.02.003. Epub 2022 Mar 11. PMID 35288066
- [Derived] Bajorin DF, Witjes JA, Gschwend JE, Schenker M, Valderrama BP, Tomita Y, Bamias A, Lebret T, Shariat SF, Park SH, Ye D, Agerbaek M, Enting D, McDermott R, Gajate P, Peer A, Milowsky MI, Nosov A, Neif Antonio J Jr, Tupikowski K, Toms L, Fischer BS, Qureshi A, Collette S, Unsal-Kacmaz K, Broughton E, Zardavas D, Koon HB, Galsky MD. Adjuvant Nivolumab versus Placebo in Muscle-Invasive Urothelial Carcinoma. N Engl J Med. 2021 Jun 3;384(22):2102-2114. doi: 10.1056/NEJMoa2034442. PMID 34077643
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT02632409.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 709 Participants Randomized, 699 Treated
Groups:
- Placebo: Placebo
- Nivolumab: Nivolumab 240mg IV Q2W
Period: Randomized
Arm/Group | Placebo | Nivolumab
Started (= Randomized) | 356 | 353
Completed (= Treated) | 348 | 351
Not Completed | 8 | 2
Not completed — AE unrelated to study Drug | 0 | 1
Not completed — Participant withdrew consent | 2 | 1
Not completed — No Longer meets study criteria | 5 | 0
Not completed — other reasons | 1 | 0
Period: Treatment Period
Arm/Group | Placebo | Nivolumab
Started (= Randomized and Treated) | 348 | 351
Completed | 132 | 143
Not Completed | 216 | 208
Not completed — Ongoing Treatment | 20 | 21
Not completed — Disease Recurrence | 147 | 90
Not completed — Study Drug Toxicity | 8 | 49
Not completed — Death | 1 | 0
Not completed — AE unrelated to study drug | 15 | 16
Not completed — Request to discontinue treatment | 4 | 19
Not completed — Participant withdrew consent | 7 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Maximum clinical benefit | 1 | 0
Not completed — No longer meets study criteria | 3 | 0
Not completed — Administrative Reason by sponsor | 0 | 1
Not completed — Other Reasons | 10 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nivolumab | Total
Number analyzed (Participants) | 356 | 353 | 709
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (8.9) | 65.3 (10.1) | 65.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 88 | 169
  Male | 275 | 265 | 540
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 16 | 37
  Not Hispanic or Latino | 143 | 142 | 285
  Unknown or Not Reported | 192 | 195 | 387
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 75 | 80 | 155
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 272 | 264 | 536
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: The time between the date of randomization and the date of first documented recurrence (local urothelial tract, local non-urothelial tract or distant), or death due to any cause, whichever occurs first.
Time Frame: approximately up to 48 months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Nivolumab
Number analyzed (Participants) | 356 | 353
Months | 10.84 [8.25 to 13.86] | 20.76 [16.49 to 27.63]
Statistical Analysis 1: Comparison: Placebo vs Nivolumab; Test type: Superiority; p = 0.0008, Stratified Cox Proportional hazard model; Hazard Ratio (HR) = 0.70, 98.22% CI 2-sided [0.55 to 0.90]

2. Primary Outcome: Disease Free Survival (DFS) in PD-L1 Expression ≥ 1% Population
Description: as for outcome 1
Time Frame: approximately up to 48 months
Population: All Randomized Participants with PD-L1 expression ≥ 1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Nivolumab
Number analyzed (Participants) | 142 | 140
Months | 8.41 [5.59 to 21.19] | NA [22.01 to NA] — Insufficient number of events to calculate median value. Upper limit number not reached
Statistical Analysis 1: Comparison: Placebo vs Nivolumab; Test type: Superiority; p = 0.0005, Stratified Cox Proportional hazard model; Hazard Ratio (HR) = 0.54, 98.72% CI 2-sided [0.35 to 0.84]

3. Secondary Outcome: Non-Urothelial Tract Recurrence Free Survival
Description: The time between the date of randomization and the date of first documented recurrence (local non-urothelial tract or distant), or death due to any cause, whichever occurs first.
Time Frame: up to 53 months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Nivolumab
Number analyzed (Participants) | 356 | 353
Months | 13.70 [8.41 to 20.34] | 22.93 [19.15 to 33.41]

4. Secondary Outcome: Non-Urothelial Tract Recurrence Free Survival in PD-L1 Expression ≥ 1% Population
Description: as for outcome 3
Time Frame: up to 53 months
Population: All Randomized Participants with PD-L1 expression ≥ 1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Nivolumab
Number analyzed (Participants) | 142 | 140
Months | 10.84 [5.65 to 22.14] | NA [24.57 to NA] — Insufficient number of events to calculate median value. Upper limit number not reached

5. Secondary Outcome: Overall Survival
Description: the time from randomization to the date of death from any cause.
Time Frame: on going
Reporting Status: Not Posted, anticipated posting 2026-01

6. Secondary Outcome: Overall Survival in Participants With PD-L1 Expression ≥ 1%
Description: the time from randomization to the date of death from any cause.
Time Frame: on going
Reporting Status: Not Posted, anticipated posting 2026-01

7. Secondary Outcome: Disease Specific Survival
Description: the time from randomization to the date of death due to disease (urothelial cancer).
Time Frame: on going
Reporting Status: Not Posted, anticipated posting 2026-01

8. Secondary Outcome: Disease Specific Survival in Participants With PD-L1 Expression ≥ 1%
Description: the time from randomization to the date of death due to disease (urothelial cancer).
Time Frame: on going
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: appoximately up to 55 months
Description: All Treated Participants
  All cause mortality is currently blinded at this time and will not be reported.
Arm/Group | Placebo | Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 129/348 | 122/351
Other Adverse Events (participants affected / at risk) | 307/348 | 332/351
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=348) | Nivolumab (N=351)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 3
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 4
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enterocele (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 0 | 2
Necrotising oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Pouchitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site extravasation (General disorders) | 0 | 1
Complication associated with device (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Sudden death (General disorders) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 2
Bronchiolitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Chest wall abscess (Infections and infestations) | 0 | 1
Citrobacter sepsis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Penile infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 5 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 5
Septic encephalopathy (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 21 | 12
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 9 | 3
Wound infection (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypobarism (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Clostridium test positive (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 | 15
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary tract carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Demyelination (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 6
Autoimmune nephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 5 | 3
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic rupture (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=348) | Nivolumab (N=351)
Anaemia (Blood and lymphatic system disorders) | 41 | 53
Hyperthyroidism (Endocrine disorders) | 4 | 37
Hypothyroidism (Endocrine disorders) | 9 | 41
Abdominal pain (Gastrointestinal disorders) | 42 | 37
Constipation (Gastrointestinal disorders) | 57 | 50
Diarrhoea (Gastrointestinal disorders) | 92 | 105
Dry mouth (Gastrointestinal disorders) | 2 | 20
Nausea (Gastrointestinal disorders) | 52 | 63
Vomiting (Gastrointestinal disorders) | 31 | 31
Asthenia (General disorders) | 31 | 42
Fatigue (General disorders) | 89 | 99
Oedema peripheral (General disorders) | 26 | 32
Pyrexia (General disorders) | 40 | 37
Nasopharyngitis (Infections and infestations) | 25 | 23
Upper respiratory tract infection (Infections and infestations) | 26 | 31
Urinary tract infection (Infections and infestations) | 55 | 68
Alanine aminotransferase increased (Investigations) | 17 | 23
Amylase increased (Investigations) | 29 | 46
Aspartate aminotransferase increased (Investigations) | 17 | 19
Blood alkaline phosphatase increased (Investigations) | 9 | 18
Blood creatinine increased (Investigations) | 49 | 51
Lipase increased (Investigations) | 30 | 40
Decreased appetite (Metabolism and nutrition disorders) | 30 | 49
Hyperglycaemia (Metabolism and nutrition disorders) | 25 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 26 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 40
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 47
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 24
Dizziness (Nervous system disorders) | 29 | 32
Headache (Nervous system disorders) | 30 | 33
Insomnia (Psychiatric disorders) | 17 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 48
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 42
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 56 | 107
Rash (Skin and subcutaneous tissue disorders) | 36 | 67
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 22
Hypertension (Vascular disorders) | 19 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT02632409/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT02632409/SAP_001.pdf